CLINICAL TRIAL: NCT07267351
Title: Determining the Effect of the ThetaHealing Meditation Method Given During the Antenatal Period on Labor Pain and Fear in Primiparous Women
Status: Enrolling by invitation | Type: Observational
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Aysenur Gezer, Research Assistant, Near East University, Turkey
Other Study IDs: EK 44/24
Record Dates: First submitted 2025-11-20; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy; Meditation; Midwifery Support; Labor Pain; Childbirth
Keywords: birth; labor pain; meditation; midwifery support
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: They are women who are between the 20th and 40th weeks of pregnancy, volunteer to participate in the study, have no systemic disease, are expected to have a normal vaginal birth, have not been diagnosed with a high-risk pregnancy, and have a singleton fetus.
  Interventions: Behavioral: ThetaHealing Meditation Method
- Experimental Group: They are women who are between the 20th and 40th weeks of pregnancy, volunteer to participate in the study, have no systemic disease, are expected to have a normal vaginal birth, have not been diagnosed with a high-risk pregnancy, and have a singleton fetus.

INTERVENTIONS:
Behavioral: ThetaHealing Meditation Method — ThetaHealing is a meditation method discovered by Vianna Stibal in 1994. This method is practiced using the theta brain wave, which has a frequency range of 4-8 Hz. According to Stibal, during the meditation process the individual has the potential to heal spiritually, physically, and emotionally (Stibal, 2011). In belief work, it actually leads the person to question what they believe and where this belief originates from, and then teaches how to load positive feelings that reflect the person's own reality in place of this negative belief. The ThetaHealing method is a defined, systematic meditation technique that is divided into courses related to various areas of life and levels of progress (Loska A., 2023).

SUMMARY:
Purpose: This randomized controlled study was designed to determine the effect of the ThetaHealing meditation method given to primiparous pregnant women during the antenatal period on labor pain and fear.

Objectives:

1. To increase childbirth satisfaction by enabling pregnant women to use the ThetaHealing meditation method during labor.
2. To ensure the use of the ThetaHealing meditation method during labor in order to reduce labor pain and/or facilitate adaptation to pain.
3. To reduce childbirth fear and/or facilitate adaptation to childbirth fear during labor by using the ThetaHealing meditation method.
4. To improve childbirth comfort through the ThetaHealing meditation method and thereby encourage vaginal birth.
5. Labor pain and childbirth fear are important factors that affect pregnant women's birth preferences. Negative birth experiences heard from women's social environment create beliefs that their own births will also be difficult, bloody, and traumatic.
6. Teaching the ThetaHealing meditation method to pregnant women during the antenatal period and enabling them to use their minds positively during labor is thought to increase women's comfort at the time of birth.

In addition, continuous midwifery care during labor is known to increase a woman's self-confidence. A woman's feeling well and safe will influence the mode of birth. There is no research in the literature specifically addressing brain waves and childbirth. However, based on information conveyed by healthcare professionals, it is thought that after the procedural processes that begin when a woman is admitted to the hospital for birth, pregnant women remain in the beta frequency together with stress and anxiety. This is because the beta frequency is a brain wave in which surrender cannot be achieved and the person experiences intense stress and anxiety. It is clear that a woman cannot reach a state of surrender while feeling anxiety and worry under bright hospital lights in a room filled with NST sounds. With the progression of labor, a calmer environment, dim lighting, and continuous midwifery support, it is thought that the pregnant woman can reach the alpha brain wave and become ready for surrender.It is even thought that if the progression of labor is left to the woman's control, she may reach the theta brain wave. A woman who can reach the alpha or theta brain wave is awake but in a continuous sleep-like state. She is now away from anxiety and stress, intuitive, instinctive, and attuned to the labor process. Since there is no scientific study on the effect of brain frequencies on the labor process, brain wave activity during labor has been inferred based on midwives' observations. By providing education on the ThetaHealing meditation method to pregnant women in the antenatal period, it is aimed to help women attune to the alpha and/or theta frequency, thereby reducing the increase in cesarean rates and facilitating adaptation to childbirth fear and pain. For these purposes, an EEG device is needed to determine in which frequency range the brain waves are during labor when the ThetaHealing meditation method is used. By investigating the effectiveness of the training using an EEG device, a contribution will be made to the literature.

DETAILED DESCRIPTION:
This randomized controlled study, planned to examine the effect of the ThetaHealing meditation method given during the antenatal period on labor pain and fear in primiparous pregnant women, is designed in three phases for the intervention group.The first phase of the study will include training of the pregnant women and implementation of the method. The training and practices will be provided only to the women in the intervention group. The training will be given to the pregnant women by the researcher in the Obstetrics and Gynecology Department of Nicosia Emergency Hospital. During the training and implementation phase, the pregnant women will attend classes once a week for four weeks, for 2 hours per day, on the predetermined day and time. The total duration of the training is planned as 8 hours. Before starting the training, the Informed Voluntary Consent Form, the Antenatal Period Information Form, and the Wijma Delivery Expectancy/Experience Questionnaire A (W-DEQ) will be administered to the couples. Visual tools, video presentations, and interactive teaching methods will be used as training materials. The exercises will be demonstrated on an individual, hands-on basis. At the end of the four-week program, the pregnant women will be given a certificate of participation and wristbands indicating that they received the training, to be worn when they come for birth. The weekly training topics and practices are presented in Appendix 7. The second phase will cover the processes of providing care and support to the pregnant woman from the onset of labor until birth. In this phase, pregnant women who have completed the training will be asked to contact the researcher when labor begins. During labor, with the support of the researcher, the pregnant woman will be guided to perform the ThetaHealing meditation method taught in the training, as well as breathing, relaxation, visualization, and deepening exercises. The hospital's standard vaginal birth follow-up procedure will be applied to the pregnant women. When cervical dilation is 3-4 cm, the VAS score will be obtained from the pregnant woman just before starting the meditation and recorded, then the ThetaHealing meditation method will be applied for 20 minutes and an EEG will be recorded by the researcher during the practice. After the practice, the VAS score will be asked again and recorded. When cervical dilation is 5-6 cm, the VAS score will again be obtained and recorded just before meditation, and during the subsequent 20-minute ThetaHealing meditation practice, EEG will be recorded. After the meditation applied in this second phase, the VAS score will be asked and recorded. When cervical dilation is 7-8 cm, the same procedure will be followed: the VAS score will be obtained and recorded before meditation, the ThetaHealing meditation method will be applied, and an EEG will be recorded by the researcher. At the end of the practice, the VAS score will be asked and recorded. During the labor process, the Visual Analog Scale (VAS) will be used, and at the end of birth the Wijma Delivery Expectancy/Experience Questionnaire B (W-DEQ) and the Postpartum Evaluation Form will be completed. Control group: The control group will consist of pregnant women from the study population who are selected by randomization and voluntarily agree to participate. The control group women who meet the sampling criteria will be informed about the study. Those who agree to participate will be given the Informed Voluntary Consent Form, the Antenatal Period Information Form, and the Wijma Delivery Expectancy/Experience Questionnaire A (W-DEQ). No additional support will be provided by the researcher to these pregnant women during pregnancy or birth. Standard delivery room care will be provided. The hospital's normal vaginal birth follow-up procedure will be applied to the pregnant women. The entire birth process of the control group will be observed by the researcher. During labor, the Visual Analog Scale (VAS) will be used, and at the end of birth the Wijma Delivery Expectancy/Experience Questionnaire B (W-DEQ) and the Postpartum Evaluation Form will be completed. The research data are planned to be collected in three phases. Phase I: For the intervention and control pregnant women who meet the study criteria, agree to participate, and are assigned by randomization, the Informed Voluntary Consent Form, the Antenatal Period Information Form, and the Wijma Delivery Expectancy/Experience Questionnaire A (W-DEQ) will be administered by the researcher. The intervention group is planned to receive a four-week, 8-hour birth preparation training in total, in the training room of the Obstetrics and Gynecology Department of Nicosia Emergency Hospital. Phase II: From the onset of labor, the pregnant women will be followed by the researcher in the delivery room. The intervention group women who participate in the study will be followed by the researcher in the standard delivery room throughout labor. For the intervention group, when cervical dilation is 3-4 cm, the breathing exercises and ThetaHealing meditation taught during the training will be applied for 20 minutes, and EEG will be recorded to determine the post-meditation frequency. The same procedure will be repeated at 5-6 cm and 7-8 cm cervical dilation, and the results will be recorded. The researcher will continue to provide support to the woman until the completion of labor. The control group women participating in the study will be followed in the standard delivery room during labor. When cervical dilation is 3-4 cm, 5-6 cm, and 7-8 cm, EEG will be recorded in three phases without applying any meditation method, and based on these EEG results, the researcher will document at which brain frequency the women are in each phase of labor without the ThetaHealing meditation method. Standard delivery room care will be provided to the pregnant women. During this process, the Visual Analog Scale (VAS) will be administered to both intervention and control group women. Phase III is planned to be conducted with the women (intervention and control) postpartum, approximately two hours after birth. The Wijma Delivery Expectancy/Experience Questionnaire B (W-DEQ) and the Postpartum Evaluation Form will be collected by the researcher through face-to-face interviews and observation.

ELIGIBILITY:
Inclusion Criteria:

A healthy pregnant woman aged between 18 and 35 years. The absence of any chronic disease. Having a single healthy fetus with a gestational age greater than 20 weeks. Willing to participate in the study. Having no systemic disease. Being in her first pregnancy.

Exclusion Criteria:

Those who do not complete the training. Not being in the 18-35 age range. Having a systemic disease. Having been diagnosed with a high-risk pregnancy. Having a multiple pregnancy. Being multiparous.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women who apply to the Obstetrics and Gynecology Outpatient Clinic and Inpatient Ward of Lefkoşa Dr. Burhan Nalbantoğlu State Hospital and agree to participate in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Determining the effect of the ThetaHealing meditation method given during the antenatal period on labor pain and childbirth fear in primiparous women. | The period from the 20th week of pregnancy until the end of labor.

CONTACTS AND LOCATIONS:
Locations (1):
- Lefkoşa Dr. Burhan Nalbantoğlu State Hospital, Nicosia, Cyprus